CLINICAL TRIAL: NCT06719921
Title: Efficacy and Safety of Catheter Ablation for Atrial Fibrillation in Non-Fluoroscopic Cardiac Electrophysiology Lab: A Non-Inferior, Multi-Center, Prospective Randomized Controlled Trial
Brief Title: Catheter Ablation for Atrial Fibrillation in Non-Fluoroscopic Lab
Acronym: NON-FLUORO-AF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Chenyang Jiang, Director of Atrial Fibrillation Center, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRRSH-2025-Research-0052
Record Dates: First submitted 2024-11-26; First posted 2024-12-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF)
Keywords: non-fluoroscopic lab; catheter ablation; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Fluoroscopic Lab Group (Experimental): Ablation procedures will utilize ICE and 3D mapping systems for non-fluoroscopic guidance. ICE is mandatory for real-time anatomical visualization.
  Interventions: Procedure: AF ablation; Other: AF ablation in a non-fluoroscopic EP lab
- Fluoroscopic Lab Group (Active Comparator): Ablation procedures will be conducted in a fluoroscopic lab. The use of ICE, 3D EP mapping systems, and other tools will follow the same recommendations as in the non-fluoroscopic lab group. Radiation exposure will be closely monitored and minimized in accordance with the ALARA (As Low As Reasonably Achievable) principles when necessary.
  Interventions: Procedure: AF ablation; Other: AF ablation in a fluoroscopic lab

INTERVENTIONS:
Procedure: AF ablation — The primary ablation strategy for both groups will be pulmonary vein isolation (PVI).
  Other additional ablation, including but not limited to linear ablation, complex fractionated atrial electrogram (CFAE) ablation, or superior vena cava (SVC) isolation is not recommended unless necessitated by one of the following:
  * Documented atrial flutter (AFL) or atrial tachycardia (AT) observed during the procedure, or
  * Arrhythmias originating from the specific region requiring intervention.
Other: AF ablation in a non-fluoroscopic EP lab — This procedure will take place in a non-fluoroscopic lab.
  Arms: Non-Fluoroscopic Lab Group
Other: AF ablation in a fluoroscopic lab — This procedure will take place in a fluoroscopic lab.
  Arms: Fluoroscopic Lab Group

SUMMARY:
This randomized controlled trial investigates the efficacy and safety of atrial fibrillation (AF) catheter ablation performed in non-fluoroscopic electrophysiology (EP) labs compared to conventional fluoroscopic digital subtraction angiography labs. The trial hypothesizes non-inferiority in outcomes, with the added benefits of simplified lab environment. Up to 724 participants aged 18-80 with paroxysmal or persistent AF will be enrolled across 10 centers. Participants will be randomized (1:1) to undergo catheter ablation in non-fluoroscopic or fluoroscopic labs, using pulmonary vein isolation (PVI) as the primary ablation strategy. The primary endpoints are freedom from AF recurrence at 12 months and composite safety outcomes related to procedure. Secondary endpoints mainly include procedure duration, recurrence during the initial 90 days, incidence of peri-procedural complications and changes in quality-of-life forms.

DETAILED DESCRIPTION:
This study evaluates the clinical efficacy and safety of AF catheter ablation procedures in non-fluoroscopic EP labs, compared to fluoroscopy labs. Non-fluoroscopic labs rely on advanced technologies such as three-dimensional electroanatomic mapping system, intracardiac echocardiography (ICE), contact force sensing catheter and/or pulsed field ablation(PFA), etc...

Participants are randomized into two groups:

1. Non-Fluoroscopic Lab Group: Ablation procedures will utilize 3D mapping systems. ICE is mandatory for real-time anatomical visualization, and fluoroscopy is employed only in unforeseen procedural challenges to ensure patient safety.
2. Fluoroscopic Lab Group: Procedures are conducted in a fluoroscopic lab using the same tools and mapping system as non-fluoroscopic lab group, with radiation exposure monitored and minimized according to ALARA principles.

The primary efficacy endpoint assesses treatment success at 12 months, defined as freedom from AF, atrial flutter (AFL), or atrial tachycardia (AT) recurrence for more than 30 seconds, as detected by ECG or 7-day Holter. Safety endpoints include a composite of major adverse events such as stroke, tamponade, myocardial infarction, or phrenic nerve injury within 3 months post-procedure. Secondary endpoints focus on procedural metrics, recurrence during the blanking period, adverse event profiles, and changes in quality-of-life forms using the AF Effect on Quality of Life (AFQT) and the EuroQol Health-Related Quality-of-Life 3-Level (EQ-5D-3L) instruments.

Data collection involves electronic data capture (EDC) systems, with detailed peri-procedural and follow-up evaluations at 3, 6, 9, and 12 months. Each participant undergoes quality-of-life assessments, physical exams, and arrhythmia recurrence monitoring via ECG and 7-day Holter recordings.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years
2. Patients diagnosed with paroxysmal AF or persistent AF with a duration of 1 years or less, who are referred for catheter ablation.
3. Patients referred for catheter ablation as a first-time intervention (no prior catheter ablation or surgical procedures for AF).
4. The patient is able and willing to provide written informed consent.

Exclusion Criteria:

1. Patients with contraindication to anticoagulation
2. Patients with contraindication to right or left sided cardiac catheterization
3. X-ray fluoroscopy is required in the procedure, such as ablation combined with VOM ethanol ablation, epicardial ablation, LAAO, CAG, etc.
4. Serious known concomitant disease with a life expectancy of < 1 year
5. MI, CABG, or PCI within the preceding 3 months
6. Left atrial diameter >55 mm
7. LVEF<30%
8. NYHA class III or IV
9. Awaiting cardiac transplantation or other cardiac surgery within 12 months.
10. History of a documented thromboembolic event within the past 6 weeks.
11. Heart or vascular malformation that impedes catheter access or vascular puncture.
12. Current enrollment in an investigational study evaluating another device or drug.
13. Acute illness, active systemic infection, or sepsis.
14. Significant congenital anomaly or a medical problem that in the opinion of the investigator would preclude enrollment in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Estimated)
Dates: Start 2025-04-22 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Freedom from Documented AF Without Antiarrhythmic Drugs at 12 Months Post-Ablation | From enrollment to the end of treatment at 12 months
  The primary end point of the study is freedom from any documented atrial arrhythmia, including AF, atrial tachycardia or atrial flutter episodes lasting longer than 30 seconds without antiarrhythmic drugs, for 12 months after the index ablation procedure, excluding a 3-month blanking period. The continuation or reinitiation of class I or class III antiarrhythmic drugs after the 3-month post-ablation blanking period, as well as electric cardioversion or catheter ablation for any atrial arrhythmias, are considered treatment failures for the primary end point.
Incidence of Composite Procedure-Related Serious Adverse Events at 3 Months Post-Ablation | From enrollment to the end of treatment at 3 months
  The primary safety endpoint is a composite of the following prespecified procedure-related serious adverse events:
  * Major vascular complication or major bleeding within the first 7 days post procedure.
  * Development of a clinically significant pericardial effusion.
  * Transient ischemic attack.
  * Stroke.
  * Myocardial infarction.
  * Sinus node dysfunction or high-grade atrioventricular block within 30 days.
  * Severe pulmonary vein stenosis.
  * Atrial-esophageal fistula, or phrenic nerve injury within 3 months.
  * Death.

SECONDARY OUTCOMES:
Acute Success of the Procedure | From the start to the completion of the procedure.
  The acute success of the procedure is defined as the percentage of procedures achieving the intended acute procedural endpoints, including: 1) Complete PVI, as confirmed by mapping or pacing maneuvers. 2) Immediate restoration and maintenance of sinus rhythm at the end of the procedure, either spontaneously or through cardioversion.
Proportion of Intra-Procedural Conversion to Using X-ray | From the start to the completion of the procedure.
  The percentage of procedures in each group (non-fluoroscopic and conventional DSA lab) that required conversion to X-ray guidance during the ablation procedure. Conversion is defined as the use of fluoroscopy to complete any part of the procedure that could not be accomplished using the assigned guidance modality.
Proportion of Patients with Recurrence of AF During the First 90 Days Post-Ablation | from the time of ablation to 90 days post-ablation.
  he percentage of patients experiencing recurrence of AF or AFL/AT during the blanking period (90 days post-ablation).
Incidence of Peri-Procedural Complications | From the start of the procedure to 7 days post-ablation.
  The percentage of patients experiencing complications such as cardiac tamponade, stroke, or vascular complications during the peri-procedural period.
Total Procedure Duration | During the procedure.
  The total time elapsed from the moment of skin puncture to the removal of all catheters and completion of the procedure (skin-to-skin time).
Ablation Time | During the procedure.
  The total time during the procedure when energy was delivered for ablation.
Change in Quality of Life Using the AF Effect on Quality of Life (AFQT) Instrument | From enrollment to the end of treatment at 12 months
  The change in patients' self-reported quality of life related to atrial fibrillation, as measured by the AF Effect on Quality of Life (AFQT) questionnaire. And the change in patients' overall health-related quality of life, as measured by the EQ-5D-3L questionnaire.
Change in Health-Related Quality of Life Using the EuroQol Health-Related Quality-of-Life 3-Level (EQ-5D-3L) Instrument | From enrollment to the end of treatment at 12 months
  The change in patients' overall health-related quality of life, as measured by the EQ-5D-3L questionnaire.

OTHER OUTCOMES:
Sub-analysis 1: Analysis of PFA VS RFA | From enrollment to the end of treatment at 12 months
  Analysis of the primary and secondary endpoints separately for RFA and PFA. All analyses will be conducted post hoc within the predefined data structure of the parent trial. No additional procedures, study visits, or participant consent are required, as this analysis relies solely on data collected as part of routine protocol-mandated assessments.
Sub-analysis 2: Impact of blanking period definitions following PFA | From enrollment to the end of treatment at 12 months
  This sub-analysis will explore the effect of different blanking period definitions (1-month, 2-month vs 3-month) on arrhythmia-free success rates after PFA, using the same dataset and follow-up schedule as the main study.
  It is an exploratory analytical component of the main trial and does not involve separate randomization or data collection.
Sub-analysis 3: Impact of AF duration and symptom/diagnosis-to-ablation interval on ablation success | From enrollment to the end of treatment at 12 months
  This sub-analysis will explore whether different time definitions influence the interpretation of 12-month ablation success. Two analytical models will be applied using the main trial dataset without additional interventions or visits:
  * Model A (documented AF duration model): Patients will be stratified by AF type (paroxysmal vs. persistent ≤1 year) and analyzed according to documented AF duration based on the first recorded AF episode.
  * Model B (symptom/diagnosis-to-ablation interval model): Patients will be stratified according to the interval from initial symptom onset or first AF diagnosis-whichever occurs earlier-to the ablation procedure, with categories defined by the actual distribution of the study population.
  This exploratory sub-analysis compares analytical approaches only; it does not modify clinical management, affect randomization, or add data collection requirements.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The IPD collected during this study will not be made publicly available. The decision not to share IPD is based on lack of resources to support secure and compliant data sharing. The study's findings are fully presented in the manuscript, and any additional summary data can be provided upon reasonable request to the corresponding author, subject to ethical considerations and institutional policies.

DOCUMENTS (1):
  • Study Protocol (2025-11-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT06719921/Prot_000.pdf